CLINICAL TRIAL: NCT05961943
Title: Feasibility, Acceptability, and Outcomes of the "RESPONSE-2" Program in Reducing Sedentary Behavior in Patients With Peripheral Arterial Disease: A Mixed Methods Pilot Study
Brief Title: RESPONSE-2-PAD to Reduce Sedentary Time in Peripheral Arterial Disease Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute for Prevention and Cardiovascular Health, Ireland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: C.A.2970
Record Dates: First submitted 2023-07-10; First posted 2023-07-27 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Peripheral Arterial Disease; Sedentary Behavior; Sedentary Time; Peripheral Arterial Occlusive Disease
Keywords: peripheral arterial disease; sedentary lifestyle; Sitting time
MeSH Terms: conditions — Peripheral Arterial Disease; Sedentary Behavior; Peripheral Arterial Occlusive Disease 1

STUDY DESIGN:
Intervention Model Description: Study recruitment will be conducted at the vascular outpatient clinic at Galway University Hospitals (GUH), Ireland. Those who consent will then be invited to attend a baseline assessment. All participants will be provided with an activPAL accelerometer device to use for seven consecutive days. Patients will also complete the six-minute walk test (6-MWT) using timed walk application. Participants will then commence the 12-week tailored intervention to empower participants to reduce/interrupt their sedentary time. Participants will have access to an online education session via the RESPONSE-2-PAD link. The researcher will support and motivate participants to reduce/interrupt their sitting time by contacting them through phone or video coaching calls once a week, on average lasting 10-15 minutes. an activity tracker will be used as a sedentary reminder. Participants will be followed up at 12-weeks and again at six months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RESPONSE-2-PAD (Experimental): All participants will use the activPAL accelerometer to quantify sedentary time/physical activity. The 6-minute-walk test will be assessed. Participants will receive the 12 week tailored intervention (RESPONSE-2-PAD link, coaching calls and activity tracker). Participants will be followed up at 12-weeks and again at six months.
  Interventions: Behavioral: RESPONSE-2-PAD

INTERVENTIONS:
Behavioral: RESPONSE-2-PAD — The RESPONSE-2-PAD program will undergo evaluation through a pilot study includes 50 patients living with peripheral arterial disease. Participants will take part in an initial assessment which will measure their sedentary time/physical activity using activPAL and their six-minute walking distance. They will then take part in a 12-week tailored, coaching-based intervention delivered remotely. The intervention involves the use of an activity tracker (sedentary reminder) and an online structured education program coupled with coaching calls that review sedentary time and activity goals weekly. At 12-weeks all participants will be invited to a follow up assessment. Participants will also be invited to take part in a semi-structured interview to explore their views and opinions of the program and its acceptability. At six months all patients will be invited for a final follow-up measurements.

SUMMARY:
The RESPONSE-2- peripheral arterial disease (PAD) program will be implemented to modify sedentary time in patients with PAD. It is an adapted version of the RESPONSE that aims to reduce sedentary behavior in individuals with diabetes. The RESPONSE-2-PAD is a multicomponent program involves an online educational component, sedentary reminders and health coaching sessions, which are designed to modify patients' sedentary behavior.

DETAILED DESCRIPTION:
Peripheral arterial disease (PAD) affects more than 230 million patients globally. PAD is characterized by a reduction in arterial perfusion caused by atherosclerotic plaque. PAD can negatively impact a person's quality of life due to the functional limitations caused by symptoms and the possibility of losing limbs. It also increases the risk of major adverse cardiac events (MACE). Many risk factors have been identified for PAD. Recently, sedentary behavior (SB) has emerged as an important risk factor for cardiovascular disease (CVD) including PAD independent to physical activity.

Studies have reported that patients with PAD have significantly higher levels of total sedentary time (ST) compared to those without PAD. Consequently, early intervention and management strategies, including addressing sedentary behavior, are crucial to prevent unfavorable outcomes in patients with established PAD as it is possible for an individual to engage in a significant amount of moderate to vigorous physical activity and have high levels of sedentary time within the same day.

The RESPONSE-2-PAD program will be evaluated in a pilot study involving 50 patients living with peripheral arterial disease. They will be recruited through the vascular services at University Hospital Galway. Those potentially interested will be provided with an information sheet. Participants will take part in an initial assessment which will measure their sitting time, physical activity participation and their six-minute walking distance. They will then take part in a 12-week individually tailored, coaching-based intervention. This intervention will be delivered remotely. The intervention involves the use of an activity tracker(sedentary reminder) and an online structured education program coupled with coaching calls (10-15minutes) that review sitting time and activity goals weekly. At 12-weeks all participants will be invited to a follow up assessment where sitting time, activity participation and six-minute walking distance will be remeasured. Patients will also be invited to take part in a semi-structured interview to explore their views and opinions of the program and its acceptability. At six months all patients will be invited for a final follow-up measurement of their sitting time, physical activity participation and six-minute walking distance in order to evaluate longer term changes.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (≥18 years),
2. Symptomatic patients with established peripheral arterial disease. PAD is confirmed by any of the following:

   * Ankle-brachial index (ABI) of less than 0.90 in at least one lower extremity
   * Toe brachial index of less than 0.60
   * Arterial occlusive disease in one lower extremity by duplex ultrasonography, computed tomographic angiography or magnetic resonance angiography.
3. Willing and able to give informed consent.
4. Can read and speak English.

Exclusion Criteria:

1. patients with significant PAD in the form of rest pain.
2. Any impairments that severely affect mobility (e.g., wheelchair bound).
3. Cognitive impairments revealed by medical records.
4. Significant comorbid disease that would significantly impair the ability to participate in activity.
5. Pregnant / lactating females.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-09-29 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Evaluating the impact of the Multicomponent Intervention (RESPONSE-2-PAD) on sedentary time in individuals with PAD. | Participants recruited for 6 months. Sedentary time assessed at baseline, after 12-week intervention, and at 6-month follow-up. Comprehensive evaluation of sedentary behavior throughout the study.
  This study will assess sedentary time in hours at baseline. After a 12-week intervention and a 6-month follow-up, sedentary time will be reassessed using the activPAL accelerometer, as done at baseline. Data analysis will evaluate changes in sedentary time from baseline to post-intervention using statistical methods to assess the effectiveness of the multicomponent intervention.
Assessing the participant involvement in RESPONSE-2-PAD Intervention to Reduce Sedentary Time. | At the end of the 6-month follow-up period, participants will be interviewed to gather qualitative feedback.
  This study aims to evaluate the level of participant engagement in the RESPONSE-2-PAD intervention, which is designed to reduce sedentary time. Through a semi structured interview. We will assess participants' involvement, motivation, and adherence to the intervention.

SECONDARY OUTCOMES:
Assessing the change in physical activity level in individuals with PAD using a Multicomponent Intervention (RESPONSE-2-PAD). | Participants recruited for 6 months. MVPA assessed at baseline, after 12-week intervention, and at 6-month follow-up.
  Moderate to vigorous physical activity (MVPA) hours will be assessed at baseline. After the intervention period (12 weeks) and 6 months follow up will be reassessed using the activPAL accelerometer as before the intervention. Then data will be analyzed to assess the changes in MVPA from baseline to post-intervention. Statistical methods will be employed to compare pre- and post-intervention MVPA and evaluate the effectiveness of the multicomponent intervention.
Assessing the Efficacy of the RESPONSE-2-PAD Program Using the 6-Minute Walk Test (6MWT) to Improve Symptom-Free Walking Distance. | 6-Minute Walk Test (6MWT) Assessments: Baseline: Before starting the intervention Post-Intervention: At the end of the 12-week intervention period Follow-Up: 6 months after the completion of the intervention
  This study aims to evaluate the effectiveness of the RESPONSE-2-PAD program in improving symptom-free walking distance using the six-minute walking test (6MWT). The assessment will include measuring total meters scored, initial claudication distance, and absolute claudication distance in participants with peripheral arterial disease (PAD).

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Jones, Principal Investigator — University of Galway; Wael Tawfick, Study Director — University of Galway; Charlotte Edwardson, Study Chair — University of Leicester
Locations (1):
- National Institute for prevention and Cardiovascular Health, Galway, Ireland

IPD SHARING:
Plan to Share IPD: Yes
Only the relevant data will be collected and stored in Galway university hospital. The data relevant to this study will only be stored for 5 more years after the thesis is written and the research has been published in peer-reviewed journals.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available to the other researchers on request for 5 years
Access Criteria: The data will be in an encrypted file and will be stored at a secure database in Galway University Hospital. Only the coded data information will be shared.

REFERENCES:
- [Background] Bailey DP, Edwardson CL, Pappas Y, Dong F, Hewson DJ, Biddle SJH, Brierley ML, Chater AM. A randomised-controlled feasibility study of the REgulate your SItting Time (RESIT) intervention for reducing sitting time in individuals with type 2 diabetes: study protocol. Pilot Feasibility Stud. 2021 Mar 19;7(1):76. doi: 10.1186/s40814-021-00816-0. PMID 33741077
- [Background] Chastin SFM, Dontje ML, Skelton DA, Cukic I, Shaw RJ, Gill JMR, Greig CA, Gale CR, Deary IJ, Der G, Dall PM; Seniors USP team. Systematic comparative validation of self-report measures of sedentary time against an objective measure of postural sitting (activPAL). Int J Behav Nutr Phys Act. 2018 Feb 26;15(1):21. doi: 10.1186/s12966-018-0652-x. PMID 29482617
- [Background] Martin A, Fitzsimons C, Jepson R, Saunders DH, van der Ploeg HP, Teixeira PJ, Gray CM, Mutrie N; EuroFIT consortium. Interventions with potential to reduce sedentary time in adults: systematic review and meta-analysis. Br J Sports Med. 2015 Aug;49(16):1056-63. doi: 10.1136/bjsports-2014-094524. Epub 2015 Apr 23. PMID 25907181